CLINICAL TRIAL: NCT05388279
Title: A Phase I Clinical Study Evaluating the Safety ,Tolerability, Pharmacokinetics of JS012 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Clinical Study to Evaluate the Safety and Tolerability of JS012 in Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the adjustment and change of the sponsor's R&D strategy, we now plan to voluntarily terminate this clinical trial.
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS012-001-I
Record Dates: First submitted 2022-05-10; First posted 2022-05-24 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Sequential
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS012 (Experimental)
  Interventions: Drug: JS012
- JS012 combination with chemotherapy (Experimental)
  Interventions: Combination Product: JS012 combine with chemotherapy

INTERVENTIONS:
Drug: JS012 — JS012, i.v., q3w
  Arms: JS012
Combination Product: JS012 combine with chemotherapy — JS012 i.v., q3w combine with chemotherapy
  Arms: JS012 combination with chemotherapy

SUMMARY:
The purpose of this phase I clinical study was to evaluate the safety and tolerability of JS012 monotherapy and combination with chemotherapy in patients with Advanced or Metastatic Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study with full informed consent and signed written informed consent form;
2. Aged ≥18 years and ≤70 years when the subject signed the informed consent;
3. Locally advanced unresectable or metastatic malignant solid tumors diagnosed histologically ;
4. Provide past tumor samples or fresh tumor tissue biopsy samples;
5. There should be at least one measurable lesion according to RECIST V1.1 evaluation criteria;
6. The expected survival is ≥3 months;
7. The physical status score is 0 or 1 on the Eastern Oncology Collaboration (ECOG) scale;
8. Good organ function;
9. Any adverse events and/or complications resulting from prior treatment, including surgery or radiation therapy, that have been adequately resolved to level 0 or 1 (according to the NATIONAL Cancer Institute Standard for General Terminology of Adverse Events (NCI-CTCAE 5.0) or to the level specified in the inclusion criteria; Any grade of hair loss/pigmentation and other long-term toxicity caused by treatment, except those that are irreversible and do not affect study dosing/compliance and patient safety at the discretion of the investigator;
10. Within 7 days prior to the first dose, women of reproductive age must be confirmed as having a negative serum pregnancy test and consent to use effective contraception during the duration of study drug use and for 90 days after the last dose. Male patients with a female partner of reproductive age agreed to use effective contraception during the study drug use period and for 90 days after the last dose.

Exclusion Criteria:

1. A history of severe allergic reactions to other monoclonal antibodies or to any component of JS012, or to other drugs or excipients involved in the trial protocol ;
2. Prior treatment with drugs or other therapies targeting CLDN18.2;
3. Malignant tumors other than the target tumor within 5 years before the first dose (except for cured cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer, or breast ductal carcinoma in situ);
4. Pregnant or lactation female patients;
5. History of allogeneic organ transplantation or hematopoietic stem cell transplantation;
6. Presence of uncontrolled or symptomatic active central nervous system (CNS) metastases;
7. Poorly controlled pleural effusion, peritoneal effusion or pericardial effusion (thoracoabdominal drainage frequency ≥1 times/month) ;
8. Clinically significant ileus;
9. Poorly controlled tumor-related pain;
10. BMI less than 17.5 at the time of signing the informed consent, or weight loss >10% in the first 2 months (significant pleural effluents should be considered) or other indicators of severe malnutrition;
11. The following within 6 months prior to the first study dose: myocardial infarction, severe/unstable angina, NYHA class 2 or higher cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestive heart failure , hypertensive crisis, or hypertensive encephalopathy; patients with known hypertension, coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must be treated with optimal stabilization as determined by the treating physician medical plan;
12. Received a drug or treatment prohibited by the protocol prior to the first dose;
13. Serious infection (CTC AE> grade 2) occurred within 28 days before the first dose, such as severe pneumonia, bacteremia, infectious complications requiring hospitalization, etc.
14. Active infection;
15. History of autoimmune disease;
16. Idiopathic pulmonary fibrosis, drug-induced pneumonia, machine-induced pneumonia (bronchiolitis obliterans), radioactive pneumonia with clinical symptoms or requiring steroid treatment, active pneumonia, or other moderate to severe lung diseases that seriously affect lung function ;
17. Inability to swallow pills, malabsorption syndrome, or any condition that affects gastrointestinal absorption;
18. The presence of other serious physical or mental disorders or abnormal laboratory tests, or the presence of alcohol or drug abuse, may increase the risk of study participation, affect treatment compliance, or interfere with study results, as well as other patients deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT | Up to approximately 41 months from first patient in.
  The Incidence of dose-limiting toxicity（DLT）
Incidence and severity of AE | Up to approximately 41 months from first patient in.
  The incidence and severity of adverse events (AE)
Incidence and severity of SAE | Up to approximately 41 months from first patient in.
  The incidence and severity of serious adverse events (SAE)
MTD | Up to approximately 41 months from first patient in.
  Determine maximum tolerated dose (MTD, if possible)
RP2D | Up to approximately 41 months from first patient in.
  Recommended phase II dose (RP2D) for JS012 monotherapy and combination therapy

SECONDARY OUTCOMES:
Drug concentrations | Up to approximately 41 months from first patient in.
  Drug concentrations in individual subjects at different time points after dosing
Cmax | Up to approximately 41 months from first patient in.
  Peak concentration
Tmax | Up to approximately 41 months from first patient in.
  Peak time
Ctrough | Up to approximately 41 months from first patient in.
  Minimum concentration
AUC0-T | Up to approximately 41 months from first patient in.
  Area under the curve from time zero to the time of the t
AUC0-INF | Up to approximately 41 months from first patient in.
  Area under the curve from time zero to infinity
t1/2 | Up to approximately 41 months from first patient in.
  elimination half-life
CL | Up to approximately 41 months from first patient in.
  clearance
MRT | Up to approximately 41 months from first patient in.
  mean retention time
Vss | Up to approximately 41 months from first patient in.
  steady-state apparent volume of distribution (Vss) (if applicable)
Css, Max | Up to approximately 41 months from first patient in.
  steady-state peak concentration Degree (Css, Max) (if applicable)
Css, min | Up to approximately 41 months from first patient in.
  Steady state minimum observed concentration (if applicable)
AUCss | Up to approximately 41 months from first patient in.
  steady-state area under curve (AUCss) (if applicable)
Rac | Up to approximately 41 months from first patient in.
  accumulation ratio (Rac) (if applicable)
Immunogenicity | Up to approximately 41 months from first patient in.
  Incidence of anti-drug antibody (ADA) and/or neutralizing antibody (Nab), titer of ADA positive samples
ADCC | Up to 21 days from pre-dose of JS012 administration in cycle 1 for each subject in the dose escalation and dose expansion phases
  Antibody Dependent cell-mediated cytotoxicity (ADCC)
CDC | Up to 21 days from pre-dose of JS012 administration in cycle 1 for each subject in the dose escalation and dose expansion phases
  Complement dependent cytotoxicity(CDC)
ORR | Up to approximately 41 months from first patient in.
  Objective response rate (ORR) was assessed based on RECIST V1.1 criteria
DOR | Up to approximately 41 months from first patient in.
  Duration of response (DOR) was assessed based on RECIST V1.1 criteria
DCR | Up to approximately 41 months from first patient in.
  Disease control rate (DCR) was assessed based on RECIST V1.1 criteria
TTR | Up to approximately 41 months from first patient in.
  Time to response (TTR) was assessed based on RECIST V1.1 criteria
PFS | Up to approximately 41 months from first patient in.
  Progression-free survival (PFS) was assessed based on RECIST V1.1 criteria
OS | Up to approximately 41 months from first patient in.
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China